CLINICAL TRIAL: NCT04523454
Title: Contraception and Pregnancy in Diabetes Mellitus
Acronym: CAPRE-DM
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 20SM5701
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 1; Contraception
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study seeks to expand upon and update this body of work. It will explore the knowledge and understanding women with diabetes have around pregnancy and conception, as well as establish how well prepared these women are for a pregnancy. Using this data, we will develop better services to inform women with diabetes about the contraception and pregnancy, as well inform the development of pre-conception counselling services for women with diabetes. If successful, we would anticipate seeing an improvement in performance in future National Diabetes in Pregnancy audits.

DETAILED DESCRIPTION:
Worldwide, 44% of pregnancies are unplanned; in the United Kingdom 45% of pregnancies and one third of births are unplanned. If a woman wants 2 children, she will spend, on average, 5 years trying to conceive or being pregnant, and 30 years trying to prevent pregnancy.

Women with diabetes are known to have 'high-risk' pregnancies. Complications for the mother include worsening diabetic control, particularly with increased hypoglycaemia in the 1st trimester; deterioration in retinopathy and nephropathy; pre-eclampsia; birth trauma due to fetal macrosomia. For the fetus, there are increased risks of congenital abnormalities; macrosomia with resultant birth trauma including shoulder dystocia; intrauterine growth restriction; miscarriage; still birth; neonatal unit admission and neonatal death.

The National Institute of Clinical and Health Excellence (NICE) guidance (NG3) contains a number of recommendations to prepare women with diabetes for a healthy pregnancy, and recommendations to avoid a pregnancy in poorly controlled diabetes; it also has recommendations about contraception. However, the National Diabetes in Pregnancy Audit 2019 shows that seven out of eight women are not adequately prepared pre-pregnancy, and there are still increased numbers of neonatal deaths, stillbirths, congenital anomalies, large and small for gestational age babies and neonatal unit admissions, compared to pregnancies in women without diabetes.

The cause for these poor outcomes, despite the NICE guidance, needs to be understood to enable pregnancy outcomes to improve. One likely factor is poor patient knowledge about the complications associated with pregnancy. One study, undertaken in 2009, showed that only 35% of women with diabetes of reproductive age recalled having any discussion about pregnancy, and only 25% were aware of any of the risks associated with pregnancy. Another study in women with diabetes seen in an antenatal clinic showed that even if a woman was aware of the risks associated with diabetes in pregnancy, she often did not attend for pre-conception counselling and preparation. The reasons for this were multifactorial, including falling pregnant faster than expected, and pervious poor interactions with healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-50 years (reproductive age) who are not currently pregnant
* Previous diagnosis of Diabetes Mellitus

Exclusion Criteria:

* Inability to understand and write in the English language
* Unable to participate due to other factors, as assessed by the Chief Investigators
* A history of gestational diabetes but not diabetes mellitus.
* Pregnant women

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Women aged 18-50 years (reproductive age) who are not currently pregnant
Study Population: Women of reproductive age (18-50) with diabetes
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rochan Agha-Jaffar, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants: All participants were women of reproductive age with known diabetes under the care of Imperial College National Health Service (NHS) Trust who agreed to participate in the study.
Period: Overall Study
Arm/Group | Participants
Started | 96 (Women who met inclusion criteria invited to complete questionnaire)
Completed | 96 (96 women completed questionnaire by point of study completion)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: As per participant flow
Groups:
- Participants: Of the 405 women who were approached to participate, 96 women completed the questionnaire.
Arm/Group | Participants
Number analyzed (Participants) | 96
Age, Continuous [Median (Full Range); unit: years] | 33 [20 to 48]
Age, Continuous [Mean (Full Range); unit: years] | 33 [20 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 57
  Unknown or Not Reported | 39
Region of Enrollment [Number; unit: participants]
  United Kingdom | 96

OUTCOME MEASURES:

1. Primary Outcome: Number of Women 'Prepared for Pregnancy\
Description: Quantitative data - Number of women 'prepared for pregnancy - HbA1C <48mmol/mol, on folic acid, on no teratogenic medications
Time Frame: 1 hour
Population: all participants
Measure: Number; unit: participants
Groups:
- Participants 'Prepared for Pregnancy': Participants on no teratogenic medicaions, HbA1C <48mmol/l and on folic acid
Arm/Group | Participants 'Prepared for Pregnancy'
Number analyzed (Participants) | 96
participants | 3

2. Secondary Outcome: Number of Women Aware of the Importance of Good Glycaemic Control Prior to Pregnancy
Description: Quantitative - Number of women aware of the importance of good glycaemic control prior to pregnancy
Time Frame: 1 hour
Population: All participants
Measure: Count of Participants; unit: Participants
Groups:
- Participants: All participants
Arm/Group | Participants
Number analyzed (Participants) | 96
Participants | 69

3. Secondary Outcome: Number of Women Who Had Attended Pre-conception Counselling
Description: Quantitative - Number of women who had attended pre-conception counselling
Time Frame: 1 hour
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Participants
Number analyzed (Participants) | 96
Participants | 17

4. Secondary Outcome: Number of Women Aware of Risks to the Foetus in Pregnancy in Women With Diabetes
Description: Quantitative - Number of women aware of risks to the foetus in pregnancy in women with diabetes
Time Frame: 1 hour
Population: All participants
Measure: Number; unit: participants
Arm/Group | Participants
Number analyzed (Participants) | 96
participants | 89

5. Secondary Outcome: Number of Women Aware of Any Risks to the Mother in Pregnancy With Pre-gestational Diabetes
Description: Quantitative - number of women aware of any risks to the mother in pregnancy with pre-gestational diabetes
Time Frame: 1 hour
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Participants
Number analyzed (Participants) | 96
Participants | 80

ADVERSE EVENTS:
Time Frame: 10 months (i.e. through whole study period) - and reviewed every month
Description: Definitions as per website clinicaltrials.gov
Groups:
- Participants: 96 women with pre-gestational diabetes who completed a questionnaire
Arm/Group | Participants
All-Cause Mortality (participants affected / at risk) | 0/96
Serious Adverse Events (participants affected / at risk) | 0/96
Other Adverse Events (participants affected / at risk) | 0/96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/54/NCT04523454/Prot_SAP_000.pdf